CLINICAL TRIAL: NCT06378385
Title: Development and Content Validation of the Childhood Early Oral Aging Syndrome (CEOAS) Index for the Deciduous Dentition
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Other Study IDs: DevelopmentCEOAS
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Observational: Development and validation of a Childhood Early Oral Aging Syndrome index for the primary dentition as a diagnostic and epidemiological survey tool considering the current changes found in the pediatric population.
  Interventions: Behavioral: Childhood Early Oral Aging Syndrome index

INTERVENTIONS:
Behavioral: Childhood Early Oral Aging Syndrome index — Development and validation of a Childhood Early Oral Aging Syndrome index for the primary dentition as a diagnostic and epidemiological survey tool considering the current changes found in the pediatric population.

SUMMARY:
Premature, non-physiological tooth wear in childhood has numerous repercussions for oral health. This is a growing problem with multifactorial causes and associated with the current lifestyle. The aim of the present study was the development and determination of content validity of the Childhood Early Oral Aging Syndrome (CEOAS) index for the primary dentition as a diagnostic and epidemiological survey tool considering the current changes found in this population.

ELIGIBILITY:
Inclusion Criteria:

-Dental surgeons

Exclusion Criteria:

-Other healthcare professionals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dental surgeons with experience in the subject of Childhood Early Oral Aging Syndrome
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Development of CEOAS index | Immediately
  The Childhood Early Oral Aging Syndrome index will be to investigate clinical signs and symptoms related to the early loss of dental structure associated with the most prevalent enamel defects, which significantly contribute to oral aging. The clinical management of tooth wear is also addressed in CEOAS scores 1, 2 and 3. Current indices used for non-carious conditions do not enable the concomitant investigation of enamel defects, which makes the proposed index innovative and of extreme important to epidemiological surveys. Understanding the prevalence of factors that either separately or synergically accelerate the process of early aging is useful to the establishment of novel treatment strategies.
  The CEOAS index involves scores of 0 to 3 for the assessment of tooth wear and dental management, whereas scores of I, II and III are used concomitantly in cases of the presence of enamel defects, as show in Table 1

SECONDARY OUTCOMES:
Validation of CEOAS index | Immediately
  Content validation will not be performed in person. The online content validation form will be sent to the specialists with the items and criteria to be assessed (Table 1) CEOAS 0 Absence of signs CEOAS 1 Mild: Presence of clinical signs in reversible stages, without sensitivity. Such cases require follow-up.
  CEOAS 2 Moderate: Presence of advanced signs with sensitivity and compromised function. Such cases require restorative treatment and management of the sensitivity.
  CEOAS 3 Severe: Presence of severe signs with pulp involvement and the risk of the loss of the tooth. Such cases require more invasive and rehabilitative treatment.
  CEOAS I Presence of PSMH - Demarcated opacities CEOAS II Presence of PSMH - Post-eruption fractures CEOAS III Presence of fluorosis

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Metropolitana de Santos - UNIMES, Santos, São Paulo, Brazil

REFERENCES:
- [Derived] Honorio Mandetta AR, Gimenez T, Sobral APT, Spinola SG, Goncalves MLL, Soares PV, Santos EM, Imparato JCP, Horliana ACRT, Mesquita-Ferrari RA, Motta LJ, Fernandes KPS, Kalil Bussadori S. Development and content validation of the Childhood Early Oral Aging Syndrome (CEOAS) index for the deciduous dentition: Research protocol. PLoS One. 2024 Oct 25;19(10):e0310543. doi: 10.1371/journal.pone.0310543. eCollection 2024. PMID 39453950